CLINICAL TRIAL: NCT02121899
Title: LUNG CAncerREgistry: An Open Registry to Measure the Impact of Adding RNA Expression Testing (myPlan Lung Cancer) on Treatment Decisions and to Assess Disease-free Survival With Long-term Follow-up in Newly Diagnosed Early Stage Lung Adenocarcinoma Patients (LUNG CARE Registry)
Brief Title: Registry Measuring Impact of RNA Expression Testing on Treatment Decisions in Early Stage Lung Cancer and Assessing the Disease-free Survival With Long-term Follow-up (ONC006)
Acronym: ONC006
Status: Terminated | Type: Observational
Why Stopped: company decision to terminate
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: myPlan ONC006
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2015-09

CONDITIONS: Lung Cancer; NSCLC; NSCLC Adenocarcinoma
Keywords: Registry
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded (FFPE) tissue from blocks or slides of prostatic adenocarcinoma biopsies.
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry is intended to measure the effect of myPlan Lung Cancer™ test has on influencing treatment decisions of Oncologists when added to standard clinical-pathological parameters in patients with early stage NSCLC.

The sponsor is conducting two parallel registries, with one directed at Surgeons (ONC003) and the other at Oncologists (ONC006). This registry is specific to Oncologists (ONC006).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early stage non-small cell lung adenocarcinoma
* Sub-population staging (IA, IB or IIA) as judged by the standard of practice at the investigational site
* Resection of tumor within previous 2 months of enrollment
* ECOG performance of 0-2
* A minimum life expectancy of six months

Exclusion Criteria

* Previous myPlan Lung Cancer test performed
* Pre-operative radiation or chemotherapy for NSCLC
* Post-operative radiation or chemotherapy for NSCLC
* Enrollment in a separate clinical trial restricting treatment options
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recently diagnosed treatment-naïve patients with early stage NSCLC (lung adenocarcinoma)
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage change from Pre-Test treatment recommendation to Post-test treatment initiated | 3 months
  The percentage change from the recorded Pre-Test treatment recommendation by the oncologist versus the Post-Test treatment initiated.

SECONDARY OUTCOMES:
Assessment of disease free survival from resection to relapse or death | 3 years
  To estimate disease-free survival with the collection of long-term follow-up information (up to 3 years post-testing).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wenstrup, MD, Study Director — Myriad Genetic Laboratories, Inc.
Locations (1):
- Orlando, Florida, United States